CLINICAL TRIAL: NCT06054165
Title: Impact of Regional Implementation of a Clinical Pathway for ELderly Patients With pelVIc Fragility fraCtures (PELVIC); a Multicenter, Stepped-wedge Randomized Controlled Trial
Brief Title: Impact of a Clinical Pathway for Pelvic Fragility Fractures
Acronym: PELVIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Noordwest Ziekenhuisgroep (Other)
Responsible Party: Principal Investigator, Dr. Daphne van Embden, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: W22_279
Record Dates: First submitted 2023-03-21; First posted 2023-09-26 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Pelvic Bone Injury; Sacral Fracture; Pelvic Fracture; Fragility Fracture
MeSH Terms: conditions — Hip Fractures | interventions — Critical Pathways

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care (No Intervention)
- Best-practice (Active Comparator)
  Interventions: Other: Clinical pathway

INTERVENTIONS:
Other: Clinical pathway — Evidence-based and expert-opinion-based clinical pathway regarding the diagnostic and treatment strategy
  Arms: Best-practice

SUMMARY:
Patients with pelvic fragility fractures suffer from high morbidity and mortality rates. Despite the high incidence of these injuries, there is currently no regional or nationwide treatment protocol which results in a wide variety of clinical practice. New insights in treatment strategies, such as early diagnosis and minimal invasive operative treatment of these fragile patient population, has led to the development of several clinical pathways in recent literature. The aim of this study is to implement an evidence and experience-based treatment clinical pathway to improve the outcomes in this fragile patient population that currently has multifactorial risks for poor outcome.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic fragility fracture caused by low energetic trauma
* Patients presented at the emergency room or out-patient clinic of a participating hospital

Exclusion Criteria:

* Patients with high suspicion of a pelvic fracture due to a malignant tumor
* Patients who are unable to follow instructions due to severe cognitive decline (for example due to dementia or Alzheimer's disease)
* Patients who pre-trauma received palliative or terminal care
* Patients who pre-trauma were wheelchair bound or bedridden
* Patients who suffer from complications from previous pelvic ring fixation
* Patients with insufficient comprehension of the Dutch language to be able to carry out the physiotherapy instructions for early mobilization

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Estimated)
Dates: Start 2024-01-21 (Actual); Primary Completion 2025-04-27 (Estimated); Study Completion 2027-04-27 (Estimated)

PRIMARY OUTCOMES:
Mobility, using the Parker mobility score (PMS) | Change from baseline PMS at 2 weeks, 3 months, 6 months, and 1 year
  Since there is no validated tool to measure mobility specifically after a pelvic fracture, the investigators choose to use The Parker mobility score as a primary outcome measurement. The Parker mobility score is a valid and reliable score measuring mobility in hip fracture patients. The Parker Mobility Score answers three questions, each valued 0-3 points, and is commonly used in clinical practice to monitor the mobility of geriatric patients. A score of 0-3 is considered low, 4-6 moderate, and 7-9 reflects good mobility. Furthermore, the Parker Mobility Score is a validated assessment tool for mortality in patients with reduced mobility after hip surgery.

SECONDARY OUTCOMES:
Mobility, using the Elderly mobility scale (EMS) | At 2 weeks, 3 months, and 1 year
  The Elderly Mobility Scale is a 20 point validated assessment tool to evaluate mobility specifically in elderly patients. The investigators decided, despite the fact that this tool has an element of measurement in it which makes it harder to determine the pre-injury score, to add this tool since it does a better job distinguishing between patients who are able to sit up and go from sitting to standing. The Elderly mobility scale ranges from 0-20 points, with high scores representing better outcome than low scores.
Functional performance, using the Katz Index of Independence in Activities of Daily Living (KATZ ADL) | Change from baseline KATZ ADL at 3 months and 1 year
  This index is one of the most commonly used scores to measure the functional status of elderly individuals. It assesses the activities of daily living using six questions, each valued 0 or 1. The score ranges from 0-6, and a score of 6 indicates full function while 4 indicates moderate impairment, and 2 or less indicates severe functional impairment
Quality of life, using the EuroQol (EQ-5D-5L) score | Change from baseline EQ-5D-5L at 1 year
  The EQ-5D-5L is a generic quality of life questionnaire which consists of a visual analogue scale and five questions about mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each question has three answer alternatives, with 1 indicating the optimal health state and 5 indicating severe problems. There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).
Return to home rate | Change from baseline place of residency at 6 weeks, 3 months, 6 months and 1 year
  The residencies will be grouped in 'living independently at home', 'assisted living', 'nursing home', 'rehabilitation centre', 'palliative care facility'.
Level of pain, using the Numerical Pain Rating Scale (NRS) | Baseline, one day post-operative (if patient underwent surgery), at 2 weeks, 6 weeks, 3 months and 1 year
  The Numerical Pain Rating Scale is an aspecific measurement tool from 0-10, with 0 reflecting no pain, 1-4 mild pain, 5-7 moderate pain, and 7-10 severe pain. This tool is currently already used by nurses in all hospitals in the Netherlands.
Descriptive name and dosage of analgesic medications used | Baseline, 2 weeks, 6 weeks, 3 months, and 1 year
  All analgesic medication that the patient is given will be recorded, and compared to the analgesic medication that the patient used prior to injury. The medication will be categorized according to the World Health Organisation analgesic ladder to facilitate comparison of changes in patients' analgesic medication usage.
Number of falls after treatment, resulting in additional injury or without injury | At 6 weeks and 3 months
  The investigators will differentiate between 'serious falls', defined as falls where the patient gets injured, and 'minor falls' where the patient did not get injured. The investigators will ask the patients during follow-up at the out-patient clinic if they fell since the last visit. The frequency of falling is related to an increased risk of mortality in elderly patients.
Number of participants with (fracture related) complications | At 2 weeks, 3 months, 6 months, and 1 year
  This includes general complications tot may occur during a period of reduced mobility or hospital admission (such as pneumonia, urinary tract infection, thromboembolic event, heart failure, cerebrovascular event, myocardial infarction). Complications related to operative treatment will also be recorded. These complications include but are not limited to: re-operation, delayed operation, infection, screw back out, malposition of screw, neurological damage. All complications will be categorized for level of severity and the necessity for further treatment according to the Clavien-Dindo classification
1-year mortality | At 1 year
  Including (presumed) cause of death
2-year mortality | At 2 year
  Including (presumed) cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Frank W Bloemers, prof, Principal Investigator — Amsterdam UMC
Locations (8):
- Netherlands (8):
  - Flevoziekenhuis, Almere Stad, Flevoland
  - Noordwest Ziekenhuisgroep, Alkmaar, North Holland
  - BovenIJ ziekenhuis, Amsterdam, North Holland
  - OLVG, Amsterdam, North Holland
  - Amsterdam UMC, Amsterdam, North Holland
  - Spaarne Gasthuis, Haarlem, North Holland
  - Dijklander Ziekenhuis, Hoorn, North Holland
  - Zaans Medisch Centrum, Zaandam, North Holland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose

REFERENCES:
- [Derived] Mennen AHM, Lommerse M, Hemke R, Willems HC, Maas M, Bloemers FW, Ponsen KJ, Van Embden D. Does regional implementation of a clinical pathway for older adult patients with pelvic fragility fractures after low-energy trauma improve patient outcomes (PELVIC): a multicentre, stepped-wedge, randomised controlled trial. BMJ Open. 2024 Aug 13;14(8):e083809. doi: 10.1136/bmjopen-2023-083809. PMID 39142675